CLINICAL TRIAL: NCT02807090
Title: Effect of Lumbar Stabilization Exercises and Circular Dances in Chronic Non Specific Low Back Pain in Middle-aged Women: Single-blind Randomized Clinical Trial
Brief Title: Effect of Lumbar Stabilization Exercises and Circular Dances in Chronic Non Specific Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: Federal University of Paraíba (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ELSE
Record Dates: First submitted 2016-05-18; First posted 2016-06-21 (Estimated); Last update posted 2019-08-06 (Actual); Status verified 2019-04

CONDITIONS: Low Back Pain
Keywords: Low Back Pain; Exercise; Dance Therapy; Physical Therapy
MeSH Terms: conditions — Low Back Pain; Motor Activity

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lumbar Stabilization Exercise (Experimental): There will be 16 sessions, twice a week, with 40-60 minutes each session. In this arm the participants will learn basic notions about anatomy and biomechanics and the lumbar stabilization technique. They will be evaluated by a pressure biofeedback in the first day that will be used in the training. The lumbar stabilization technique consists of three stages: cognitive, associated and automatic. The biofeedback is used in the first stage and it helps patients to do the best contraction of stabilization muscles in different levels of pressure. Then, in stage two the patients do the contraction without the use of biofeedback and in the last phase different exercises are associated with the contraction of stabilization muscles.
  Interventions: Other: Lumbar Stabilization Exercise
- Circular Dance (Experimental): There will be 16 sessions, twice a week, with 60 minutes each session. In this arm the participants will do the exercises in a group of 20 subjects. In every meeting there will be the follow stages: reception, reflection, warming/stretching, explanation about circular dance, choreography orientation, practice and finishing.
  Interventions: Other: Circular dance

INTERVENTIONS:
Other: Lumbar Stabilization Exercise — There will be 16 sessions, twice a week, with 40-60 minutes each session. In this arm the participants will learn basic notions about anatomy and biomechanics and the lumbar stabilization technique. They will be evaluated by a pressure biofeedback in the first day that will be used in the training. The lumbar stabilization technique consists of three stages: cognitive, associated and automatic. The biofeedback is used in the first stage and it helps patients to do the best contraction of stabilization muscles in different levels of pressure. Then, in stage two the patients do the contraction without the use of biofeedback and in the last phase different exercises are associated with the contraction of stabilization muscles.
  Arms: Lumbar Stabilization Exercise
Other: Circular dance — There will be 16 sessions, twice a week, with 60 minutes each session. In this arm the participants will do the exercises in a group of 20 subjects. In every meeting there will be the follow stages: reception, reflection, warming/stretching, explanation about circular dance, choreography orientation, practice and finishing.
  Arms: Circular Dance

SUMMARY:
Supervised exercises are the first line therapy for patients with chronic low back pain. The lumbar segmental stabilization (LSE) is a specific training for the muscles of the lumbar spine, which aims to improve neuromuscular control, strength and endurance of the muscles that promotes stability to the spine. The circular dance (CD) belongs to the group of complementary and integrative practices entered in Public Health Care in Brazil, and has been used to improve several aspects related to physical and mental states such as flexibility, posture, strength and muscular endurance, awareness or scheme body, pain control and strains. There are few studies evaluating the circular dance effect on back pain. The aim of this study is to compare the effects of lumbar stabilization exercises and circular dance for improvement in non specific low back pain in middle-aged women.

DETAILED DESCRIPTION:
OBJECTIVE: To compare the effect of CD with ESL exercises on pain and functional disability in women with nonspecific chronic low back pain (DLCI). METHOD: Thirty-eight women, aged 35-60 years, were randomly assigned to two groups: 1) Circular Dance group (gDC); 2) Lumbar Stabilization Exercise group (gESL). The primary clinical outcomes were pain, assessed using the Numerical Pain Scale and functional disability by the Roland Morris Disability Questionnaire and the secondary outcomes were: Depression assessed by the Beck Depression Inventory; Anxiety by the Numerical Anxiety Scale; Global Perception with the Global Effect Perception Scale, Signs and Symptoms of Adverse Effects analyzed by the Collective Subject Discourse and Quality of Life method using the Short-Form Health Survey Questionnaire (SF-36). The groups were treated twice a week for 60 minutes for 8 weeks totaling 16 sessions. Each participant was assessed before and after treatment and at follow-up 12 and 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Diagnose of non specific low back pain for a period of three months without radiculopathy symptoms
* Seek treatment

Exclusion Criteria:

* Inflammatory disorders of the spine
* Spinal tumors
* Spine surgery
* Unconsolidated fractures or malunion of the spine
* Rheumatologic disease
* Spondylolysis or spondylolisthesis
* Patients who are in labor dispute
* Patients undergoing physical therapy or drug treatment to opioid-based

Ages: 35 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2018-07 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
Change in pain through Pain visual analogue scale | Before the treatment and after the treatment (immediately after the treatment, and 4 and 16 weeks after treatment) and in every session (from the first session to the sixteen session), immediately after session
  Scale with 11 centimeters is used for evaluate pain intensity

SECONDARY OUTCOMES:
Roland Morris Disability Questionnaire | Before and after the treatment (immediately after the treatment, and 4 and 16 weeks after treatment)
  This questionnaire evaluate the functional disability provoked by Low back pain
Global Perceived Effect Scale | Before and after the treatment (immediately after the treatment, and 4 and 16 weeks after treatment)
  This scale evaluates the participant's perception of recovery from the treatment, comparing the symptoms at the beginning and at the end of treatment.
Beck Depression Inventory | Before and after the treatment (immediately after the treatment, and 4 and 16 weeks after treatment)
  Composed of 21 items, this scale evaluates the intensity of symptoms and ranges from 0 to 3 and the higher the score, the greater the depressive symptoms.
Visual analogue scale for anxiety | Before and after the treatment (immediately after the treatment, and 4 and 16 weeks after treatment)
  Scale of 11 points, whose value ¨0¨ in the left end indicates ¨ without anxiety¨ and the value ¨10¨ in the extreme right indicates "the worst perceived anxiety" in the last seven days
Medical Outcomes Study 36 - Item Short - Form Health Survey | Before and after the treatment (immediately after the treatment, and 4 and 16 weeks after treatment)
  This instrument evaluates the patient's perception of his quality of life in aspects related to functional capacity, physical aspects, pain, general health, vitality, social, emotional and mental health aspects.
Symptoms and Adverse events or side effects | Before and after the treatment (immediately after the treatment, and 4 and 16 weeks after treatment)
  During treatment, patients are asked about side effects resulting from the treatment performed.

CONTACTS AND LOCATIONS:
Overall Officials: Raquel A Casarotto, PhD, Study Director — University of Sao Paulo
Locations (1):
- Juerila Moreira Barreto, João Pessoa, Paraíba, Brazil

IPD SHARING:
Plan to Share IPD: No